CLINICAL TRIAL: NCT01329250
Title: Pharmacokinetics and Safety of Moxifloxacin; a Dose Escalation in Patients With Tuberculosis
Brief Title: Pharmacokinetics and Safety of Moxifloxacin
Acronym: MFX468
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow enrolment of patients and new insights
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, JWC Alffenaar, PharmD, PhD, University Medical Center Groningen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MFX468
Record Dates: First submitted 2011-03-08; First posted 2011-04-05 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Moxifloxacin; Pharmacokinetics; Safety
MeSH Terms: conditions — Tuberculosis | interventions — Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Moxifloxacin (Experimental): Moxifloxacinin escalating dose
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Moxifloxacin — Patients will start on a standard dose of MFX 400 mg once daily. After 8 days the dose will be increased to 600 mg once daily and on the 15th day of treatment, the dose of MFX will be escalated to 800 mg. In patients who have been treated with rifampicin (RIF) in the past three weeks prior to start of MFX treatment an additional washout period of 3 weeks to reduce the rifampicin induced enzymatic activity will precede the dose escalation.
  Other Names: MFX

SUMMARY:
The main objective of this prospective clinical trial is to compare pharmacokinetics and safety and tolerability of a standard dose (400 mg) with an escalated dose (600 mg; 800 mg) of moxifloxacin (MFX). This clinical trial will provide important safety information on MFX in a higher dosage in TB patients.

DETAILED DESCRIPTION:
Moxifloxacin (MFX) is a fluoroquinolone with a high in vitro and in vivo bactericidal activity against Mycobacterium tuberculosis. A daily dose of 600-800 mg MFX should be considered for optimal killing of the involved mycobacteria and suppression of drug resistance, which is higher than the currently used dose of 400 mg once daily. In general, safety data to support switching to the suggested higher dose are limited.

For this purpose, twenty tuberculosis patients will start on a standard dose of MFX 400 mg once daily. After 8 days the dose will be increased to 600 mg once daily and on the 15th day of treatment, the dose of MFX will be escalated to 800 mg. In patients who have been treated with rifampicin (RIF) in the past three weeks prior to start of MFX treatment an additional washout period of 3 weeks to reduce the rifampicin induced enzymatic activity will precede the dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with TB, with Mycobacterium tuberculosis (or M. africanum) by culture
* Starting treatment with MFX in a dose of 400 mg as part of their TB treatment

Exclusion Criteria:

* Contra-indication for MFX
* Baseline QTc-interval > 450 msec
* History of resuscitation
* History of ventricular tachycardia (including Torsades de Pointes)
* Family history of sudden cardiac death or Torsades de Pointes
* Additional risk factors for Torsades de Pointes (including known heart failure, Left ventricular hypertrophy)
* Use of concomitant treatment with QT/QTc prolonging drugs (including anti-dysrhythmics class IA and III, antipsychotics, tricyclic antidepressants or the antihistaminic drug terfenadine)
* Abnormal electrolytes (K, Mg, Na, Ca)
* Abnormal cardiac repolarisation on screening/baseline ECG
* History of adverse events to fluoroquinolones
* HIV co-infection
* RIF treatment during last 3 weeks before start of the study. After a washout period of 3 weeks the patient can be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-05; Primary Completion 2015-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Bound area under the plasma concentration-time curve (AUC0-24h) relative to the minimal inhibitory concentration (MIC) | 7 days post dosage
  % of patients who will reach an AUC0-24h/MIC ratio of at least 100 after administration of 400 mg (i.e. 7 days post dosage) moxifloxacin
Unbound AUC0-24h/MIC ratio as predictive parameter for efficacy of unbound MFX dose escalated treatment of tuberculosis | 7 days post dosage
  % of patients who will reach an unbound AUC0-24h/MIC ratio of at least 60 after administration of 400 mg (i.e. 7 day post dosage) moxifloxacin.
Bound AUC0-24h/Mutant Prevention Concentration (MPC) ratio | 7 days post dosage
  % of patients who will reach an adequate AUC0-24h/MPC ratio of at least 93 after administration of 400 mg (i.e. 7 days post dosage) moxifloxacin
Unbound AUC0-24h/MPC ratio as predictive parameter for efficacy of unbound MFX dose escalated treatment of tuberculosis and suppression of MFX resistance | 7 days post dosage
  % of patients who will reach an unbound AUC0-24h/MPC ratio of at least 53 after administration of 400 mg (i.e. 7 days post dosage) moxifloxacin
% of patients having adverse effects, including QT interval prolongation, hypersensitive reactions, diarrhoea, vomiting and hepatic or renal injury | up to 21 days
  * QT interval in msec
  * Percentage of patients developing hepatic toxicity grade ≥ 2 or 3 Common Toxicity Criteria (CTC)
  * Percentage of patients developing renal toxicity grade ≥ 2 CTC
Bound area under the plasma concentration-time curve (AUC0-24h) relative to the minimal inhibitory concentration (MIC) | 14 days post dosage
  % of patients who will reach an AUC0-24h/MIC ratio of at least 100 after administration of 600 mg (i.e. 14 days post dosage) moxifloxacin
Bound area under the plasma concentration-time curve (AUC0-24h) relative to the minimal inhibitory concentration (MIC) | 21 days post dosage
  % of patients who will reach an AUC0-24h/MIC ratio of at least 100 after administration of 800 mg (i.e. 21 days post dosage) moxifloxacin
Unbound AUC0-24h/MIC ratio as predictive parameter for efficacy of unbound MFX dose escalated treatment of tuberculosis | 14 days post dosage
  % of patients who will reach an unbound AUC0-24h/MIC ratio of at least 60 after administration of 600 mg (i.e. 14 days post dosage) moxifloxacin.
Unbound AUC0-24h/MIC ratio as predictive parameter for efficacy of unbound MFX dose escalated treatment of tuberculosis | 21 days post dosage
  % of patients who will reach an unbound AUC0-24h/MIC ratio of at least 60 after administration of 800 mg (21 days post dosage) moxifloxacin.
Bound AUC0-24h/Mutant Prevention Concentration (MPC) ratio | 14 post dosage
  % of patients who will reach an adequate AUC0-24h/MPC ratio of at least 93 after administration of 600 mg (i.e. 14 days post dosage) moxifloxacin
Bound AUC0-24h/Mutant Prevention Concentration (MPC) ratio | 21 post dosage
  % of patients who will reach an adequate AUC0-24h/MPC ratio of at least 93 after administration of 800 mg (i.e. 21 days post dosage) moxifloxacin
Unbound AUC0-24h/MPC ratio as predictive parameter for efficacy of unbound MFX dose escalated treatment of tuberculosis and suppression of MFX resistance | 14 days post dosage
  % of patients who will reach an unbound AUC0-24h/MPC ratio of at least 53 after administration of 600 mg (i.e. 14 days post dosage) and moxifloxacin
Unbound AUC0-24h/MPC ratio as predictive parameter for efficacy of unbound MFX dose escalated treatment of tuberculosis and suppression of MFX resistance | 21 days post dosage
  % of patients who will reach an unbound AUC0-24h/MPC ratio of at least 53 after administration of 800 mg (i.e. 21 days post dosage) moxifloxacin

SECONDARY OUTCOMES:
Evaluation of the predictive performance of the limited sampling strategies based on a pharmacokinetic population model to calculate AUC0-24h. Several limited sampling points will be evaluated. | 7 days post dosage
  Several limited sampling strategies to predict moxifloxacin AUC0-24h, based on limited sampling points, will be evaluated after administration of 400 mg (i.e. 7 days post dosage)moxifloxacin
Correlation between MFX concentration (mg/L) and QT interval (msec) | 7 days post dosage
  Correlation between MFX concentration (mg/L) and QT interval (msec) after administration of 400 mg (i.e. 7 days post dosage) moxifloxacin
Correlation of drug exposure (AUC) and adverse effects | up to 21 days
  * vomiting and diarrhoea
  * QT interval (msec)
Correlation between the genetic risk score and MFX induced QT prolongation | up to 21 days
Evaluation of the predictive performance of the limited sampling strategies based on a pharmacokinetic population model to calculate AUC0-24h. Several limited sampling points will be evaluated. | 14 days post dosage
  Several limited sampling strategies to predict moxifloxacin AUC0-24h, based on limited sampling points, will be evaluated after administration of 600 mg (i.e. 14 days post dosage) moxifloxacin
Evaluation of the predictive performance of the limited sampling strategies based on a pharmacokinetic population model to calculate AUC0-24h. Several limited sampling points will be evaluated. | 21 days post dosage
  Several limited sampling strategies to predict moxifloxacin AUC0-24h, based on limited sampling points, will be evaluated after administration of 800 mg (i.e. 21 days post dosage) moxifloxacin
Correlation between MFX concentration (mg/L) and QT interval (msec) | 14 days post dosage
  Correlation between MFX concentration (mg/L) and QT interval (msec) after administration of 600 mg (i.e. 14 days post dosage) moxifloxacin
Correlation between MFX concentration (mg/L) and QT interval (msec) | 21 days post dosage
  Correlation between MFX concentration (mg/L) and QT interval (msec) after administration of 800 mg (i.e. 21 days post dosage) moxifloxacin

CONTACTS AND LOCATIONS:
Overall Officials: Jos GW Kosterink, PharmD, PhD, Study Chair — Univeristy Medical Center Groningen; Jan-Willem C Alffenaar, PharmD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands